CLINICAL TRIAL: NCT04921124
Title: Pharmacokinetic and PHarmacodynamic Analysis and Evaluation of Teriparatide (PTH 1-34) Between Sexes
Acronym: PHAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other); Ministry of Defence, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHAB01
Record Dates: First submitted 2021-05-19; First posted 2021-06-10 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Stress Fracture
MeSH Terms: conditions — Fractures, Stress | interventions — Teriparatide

STUDY DESIGN:
Intervention Model Description: This is an open-label, parallel, clinical trial in two separate groups, men and women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Teriparatide, 20 µg Subcutaneous (S/C) per day.
  Two doses in total.
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — PTH(1-34) cartridge and pen device

SUMMARY:
To test for a difference in the pharmacokinetics (PK) and pharmacodynamics (PD) of teriparatide (PTH 1-34), between healthy male and female volunteers matched to military recruits in training.

DETAILED DESCRIPTION:
Teriparatide, first licensed for fracture prevention in osteoporosis in 2003, is a human recombinant preparation of parathyroid hormone (PTH) 1-34. The licensed dose is a 20 µg sub-cutaneous (S/C) injection delivered once daily using a pre-filled pen. Published pharmacokinetic (PK) and pharmacodynamic (PD) data focus on administration in adult female pre-menopausal women. Eli Lilly did not publish their original 'First in Human' data, therefore there is a lack of available data in men. The patent on the Eli Lilly formulation expired in August 2019 and three teriparatide biosimilars have been released onto the UK market. Gedeon Richter and Thornton and Ross presented data in osteoporotic patients to the MHRA to license their products as biosimilars. Teriparatide has also been investigated in the treatment of stress fractures, but there are no published data comparing the PKs and PDs of these drugs in a population equivalent to individuals undergoing military training (i.e. young healthy men and women).

Existing data to support the equivalence of teriparatide between sexes is limited. Citrate and calcium infusions have been used to characterise the impact of sex differences on PTH dynamics in twelve women with mean age ± SD of 26.4 ± 1.6 years and 12 men with mean age of 26.6 ± 1.3 years. They reported no between sex differences in serum PTH concentrations. It has also been reported that 2-weeks of intermittent PTH administration in mice was anabolic for cortical bone, with a greater effect observed in male compared with female animals. No studies have investigated between sex PK or PD differences or efficacy of teriparatide injection in humans. By examining this, the present study will help to further our understanding of how teriparatide can be used in men and women.

A review considering a number of trials supported the use of PTH in its licensed indications and demonstrated the efficacy of this drug in both male and female subjects. The evidence base cited in this review is primarily from post-menopausal women in line with the licensed indication.

This study compliments the RETURN trial which is investigating the efficacy of teriparatide for accelerating stress fracture healing in Army infantry recruits (EudraCT: 2018-002130-20). The study is based at the Infantry Training Centre (ITC), which currently predominantly trains men, hence men will form the majority of the RETURN study participants. Opening front line roles to women comes with a well-documented risk of musculoskeletal injury due to the nature of infantry training (HQ Army, 2016). If the results of the RETURN trial are to be extrapolated to women and inform Defence treatment policy for stress fractures, the between sex differences in PK and PD in a population matched to individuals in military training must be established. This study is required if the results of RETURN are to be extrapolated to a female population undergoing military training.

The Gedeon Richter preparation, 'Terossa' will be used in this study as this is the preparation that is being used in the RETURN study. This will control for inter-brand variation.

Nephrogenous cyclic Adenosine Mono Phosphate is a measurement of PTH 1-34 activity at the kidney and can therefore be used to estimate the early biological effects of PTH 1-34 in humans.

The research questions are;

1. Is there a difference in the PK or PD profile of teriparatide subcutaneous injection between men and women?
2. Are the PK and PD measurements reliable and reproducible? The cohort for investigation is young healthy (free from immune, cardiovascular or metabolic diseases) men and women, military or physically trained civilians, free from illness, and matched to a military population in training, based on age, body mass index (BMI) and absence of medical conditions that would be a bar to entry to the Army (Can I Join The Army | Find Out if You Are Eligible | British Army - British Army Jobs (mod.uk) [Accessed 16/01/2021]).

The intervention involves a single dose of teriparatide administered on 2 occasions.

Participants will be closely monitored for 12 hours, plus a further 12 hours urine collection followed by a 24-hour washout period.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent to participate;
* Be able to comply with protocol;
* Be able to adequately understand written and spoken English;
* Be aged between 18 and 36 years;
* Have a BMI ≥18.5 and ≤28.0 kg/m2;
* Regularly perform a minimum of 3 sessions / week of 40 minutes or more of moderate or vigorous exercise;
* Be without any clinically significant illness (free from immune, cardiovascular or metabolic diseases and absence of medical conditions that would be a bar to joining the Army),
* Have baseline blood tests within reference range as per screening assessment table (table 1). Minor abnormalities will be assessed by the PI. Participants will still be eligible if these are felt to be of no clinical importance and this decision is documented by the PI;
* Be vitamin D replete (25(OH)D ≥50 nmol/L). Potential participants presenting with 25(OH)D <50 nmol/L I will be offered supplementation and may be re-screened once their course of treatment is complete

Exclusion Criteria:

* Hypersensitivity to the active PTH or any of the excipients listed in any of the SmPCs.
* Pre-existing hypercalcaemia
* Participants with skeletal malignancies or bone metastases.
* Significant musculoskeletal injury or fracture within the last 6 months. Significance to be determined by the PI.
* Digoxin and any other concurrent therapy that, in the investigators' opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Pregnancy, suspected pregnancy or breastfeeding. Female participants must have a negative urine pregnancy test at screening and be willing and able to use a medically accepted method of birth control (reliable use of oral contraceptive, hormonal intrauterine device, non-hormonal intrauterine device with condom, diaphragm with condom, or condom with spermicide) from the screening visit through to the end of the experimental testing visit or declare that they are abstaining from sexual intercourse from the screening visit through the end of the experimental testing visit or are surgically sterile (have undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
* Less than 6 months post-partum.
* Less than 6 months post-breastfeeding.
* Severe renal impairment (eGFR <30mLs/min/1.73m2).
* Pre-existing metabolic bone diseases including hyperparathyroidism and Paget's disease of the bone.
* Unexplained elevations of total ALP.
* Prior external beam or implant radiation therapy to the skeleton.
* Participating in a concurrent drug trial. Potential participants will be excluded if they have been in receipt of an investigational drug or biological agent within the last 4 weeks (or 5 times the half-life if this is longer) prior to study entry.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Concentration over time assessed by the area under the curve (AUC) of teriparatide (PTH (1-34)). | One dose (24 hours)
  Compared in men and women.
The maximum concentration (Cmax) for teriparatide (PTH 1-34). | One dose (24 hours)
  Compared in men and women.

SECONDARY OUTCOMES:
Changes in cAMP production over time following a single dose of teriparatide. | One dose (24 hours)
  Compared in men and women.
Changes in cAMP metabolism over time following a single dose of teriparatide. | One dose (24 hours)
  Compared in men and women.
The reproducibility of Concentration over time assessed by the area under the curve (AUC) of teriparatide (PTH (1-34)). | Two doses (24 hours wash out between )
  Compared in men and women.
The reproducibility of changes in cAMP production over time following a repeated dose of teriparatide. | Two doses (24 hours wash out between )
  Compared in men and women.
The reproducibility of changes in cAMP metabolism over time following a repeated dose of teriparatide. | Two doses (24 hours wash out between )
  Compared in men and women.

CONTACTS AND LOCATIONS:
Overall Officials: William Fraser, Prof, Principal Investigator — UEA
Locations (1):
- Norfolk and Norwich University Hospitals Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No